CLINICAL TRIAL: NCT03853681
Title: Study on the Response to Tetanus Vaccination of People Living With HIV
Acronym: VACTEVIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Niort (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PI-2019-02
Record Dates: First submitted 2019-02-15; First posted 2019-02-26 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- additional blood sampling (Other)
  Interventions: Diagnostic Test: additional blood sampling

INTERVENTIONS:
Diagnostic Test: additional blood sampling — additional blood sampling

SUMMARY:
The response to primary tetanus immunization of HIV-infected children is lower than that of uninfected children.

Response to tetanus toxoid (TT) booster doses in adults living with HIV who have received primary vaccination prior to infection is not known.

Currently, it is recommended to have a TT booster for people living with HIV (PLHIV) every 10 years. In general population, this recall is made only at 25, 45 and 65 years, then every 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Person aged ≥ 18 years
* Person infected with HIV followed in the infectious diseases department of CH Niort
* Born in France
* Affiliate or beneficiary of a social security scheme
* Being able to give free and informed consent to participation in research

Exclusion Criteria:

* Persons with a contraindication to tetanus vaccination
* Persons under guardianship or curatorship or without civil law

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
the vaccine response to tetanus vaccination | Month 6
  An anti-tetanus IgG level> 0.1 is considered long-term protective. An anti-tetanus IgG level between 0.01 and 0.1 is considered protective in the short term.
  The measurement of the vaccine response will be correlated with the age of the last VAT recall (<10 years, between 10 and 20 years,> 20 years and unknown)

CONTACTS AND LOCATIONS:
Overall Officials: Simon SUNDER, Doctor, Study Director — Centre Hospitalier de Niort - France; Simon SUNDER, Doctor, Study Director — CH Niort
Locations (1):
- Centre Hospitalier de Niort, Niort, France

IPD SHARING:
Plan to Share IPD: No